CLINICAL TRIAL: NCT01165307
Title: A Prospective Randomized Trial of Medical Therapy Versus Radiofrequency Endometrial Ablation in the Initial Treatment of Menorrhagia: Treatment Outcomes and Cost Utility Analysis
Brief Title: Medical Therapy Versus Radiofrequency Endometrial Ablation in the Initial Treatment of Menorrhagia
Acronym: iTOM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abimbola Famuyide (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Abimbola Famuyide, Consultant, Assistant Professor of Obstetrics-Gynecology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-007334
Record Dates: First submitted 2010-07-09; First posted 2010-07-19 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; Endometrial ablation; Heavy menstrual bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Estradiol; Levonorgestrel; Ethinyl Estradiol-Norgestrel Combination; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Therapy (Active Comparator): Subjects will be prescribed monthly packets of Estradiol 30mcg / Levonorgestrel 150mcg monophasic oral contraceptive pills. Subjects who are unable to tolerate oral contraceptive pills or are unwilling to take oral contraceptive pills will be prescribed naproxen sodium pills. The latter will be administered as follows; 500mg with onset of menses, then 250mg three times daily for the duration of the menses (or maximum of five days).
  Interventions: Drug: Estradiol 30mcg / Levonorgestrel 150mcg monophasic oral contraceptive pills; Drug: Naproxen sodium pills
- Radiofrequency Endometrial Ablation (Active Comparator): Subjects will undergo NovaSure® radiofrequency endometrial ablation within 4 weeks of randomization. The procedure will occur at any time during the menstrual cycle, without endometrial pre-treatment. Endometrial thinning will be carried out using suction curettage in 50% of the cases included in the ablation group. Random assignment for this treatment will be included in the overall randomization plan.
  Interventions: Device: NovaSure® Radiofrequency Endometrial Ablation

INTERVENTIONS:
Drug: Estradiol 30mcg / Levonorgestrel 150mcg monophasic oral contraceptive pills — Each packet consists of a fixed dose of 30mcg estradiol and a 150mcg dose of levonorgestrel for the first 21 days of the cycle, followed by a 7 day pill free period. Subjects will be instructed to administer the pills orally, starting 5 days after the start of menstrual blood flow, continuing cyclically, thus allowing for withdrawal bleeding after the 21 day pill cycle.
  Other Names: Nordette®
  Arms: Medical Therapy
Drug: Naproxen sodium pills — As an alternative to oral contraceptive pills, subjects may take Naproxen 500 mg with onset of menses, then 250 mg three times daily for the duration of the menses (or maximum of five days)
  Other Names: Naprosyn 250 mg tablets
  Arms: Medical Therapy
Device: NovaSure® Radiofrequency Endometrial Ablation — Radiofrequency endometrial ablation is performed in the outpatient surgery department. Subjects receive intravenous medication, determined by the attending anesthesiologist, sufficient to induce conscious sedation during the procedure.
  Arms: Radiofrequency Endometrial Ablation

SUMMARY:
Excessive menstrual loss (menorrhagia) is a common condition that affects women of reproductive age, and can result in anemia, chronic fatigue and lost wages from work. The traditional first line management involves treatment with oral contraceptives or non-steroidal anti-inflammatory agents. Many women ultimately undergo hysterectomy, a major operative procedure associated with increased costs, loss of feeling of womanhood, debilitating complications and on rare occasions, death.

The newer global endometrial ablation (GEA) devices allow the destruction of the endometrial lining, without the removal of the uterus, in an ambulatory surgery setting. GEA offers a safe and effective alternative to hysterectomy with minimal risks and without unpleasant side-effects.

Presently, global endometrial ablation is offered as an alternative to hysterectomy, after medical intervention has failed. This study will determine the role of global endometrial ablation in the initial management of menorrhagia. Women seeking treatment for menorrhagia will be randomized to either the medical treatment arm or the global endometrial ablation arm.

This study will be the first to compare clinical efficacy and costs between oral contraceptive pills and global endometrial ablation in the initial management of menorrhagia and could potentially change the management of menorrhagia and impact millions of women who suffer from this condition.

DETAILED DESCRIPTION:
Goal of study: To evaluate the safety, effectiveness as well as cost- effectiveness of Global Endometrial Ablation (GEA) as an initial treatment for menorrhagia.

Specific aim #1: To determine if global endometrial ablation (GEA) is more effective than medical therapy in the initial management of menorrhagia.

Specific aim #2: To determine disease-specific resource utilization and costs associated with the treatment alternatives and the cost effectiveness of global endometrial ablation (GEA) compared with medical treatment (oral contraceptive pills) in the initial management of menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female, ages 30-55, who is pre-menopausal and for whom childbearing is complete
2. Subjective symptom of excessive menstrual loss
3. Normal uterine cavity length (≥ 4cm) with a sound measurement of ≤10cm documented by sonohysterogram or hysteroscopy in the preceding 6 months
4. At least one normal Pap Test and no unexplained abnormal Pap Tests within 6 months of procedure
5. Prior history of permanent sterilization or use of reliable non-hormonal contraception during the 14 month study period or history of vasectomy in partner
6. Freely agree to participate in the study including all study related procedures and evaluations, and document this agreement by signing the informed consent document

Exclusion Criteria:

1. Pregnancy or desire for future childbearing
2. Active lower genital infection at the time of procedure
3. Active urinary tract infection at the time of procedure
4. Active pelvic inflammatory disease (PID) or recurrent chronic PID
5. Endometrial neoplasia, determined by endometrial biopsy taken within 12 months of study entry
6. Current or past history of cervical or endometrial cancer
7. Uterine sound measurement greater than 10cm
8. Submucous leiomyoma greater than 2cm or cavity distorting leiomyoma
9. History of myomectomy or classical cesarean section
10. Previous endometrial ablation
11. Oral hormonal treatment in the preceding 3 months, hormone releasing intrauterine contraceptive in the preceding month, or injectable hormone treatment in the preceding 12 months
12. Contraindication to hormonal therapy and non-steroidal anti-inflammatory agents.
13. History of a coagulopathy or endocrinopathy
14. Inability to follow up at 12 months

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2009-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abimbola O. Famuyide, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Famuyide AO, Laughlin-Tommaso SK, Shazly SA, Hall Long K, Breitkopf DM, Weaver AL, McGree ME, El-Nashar SA, Lemens MA, Hopkins MR. Medical therapy versus radiofrequency endometrial ablation in the initial treatment of heavy menstrual bleeding (iTOM Trial): A clinical and economic analysis. PLoS One. 2017 Nov 15;12(11):e0188176. doi: 10.1371/journal.pone.0188176. eCollection 2017. PMID 29141040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota from September 2009 to February 2013.
Pre-assignment Details: 77 subjects were initially consented, but 10 subjects were not randomized because 4 declined participation after consent, 4 reported spontaneous improvement during initial evaluation, 1 had an abnormal Pap smear indicating treatment, and 1 had a polypoid mass on hysteroscopy.
Period: Overall Study
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Started | 33 | 34
Completed | 19 | 31
Not Completed | 14 | 3
Not completed — Lost to Follow-up | 11 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Subject not available for contact | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (5.5) | 41.9 (6.0) | 42.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Menstrual Blood Loss (MBL) as Measured by Pictorial Blood Loss Assessment Chart (PBLAC).
Description: The PBLAC is a simple, pictorial tool used in women with menorrhagia to assess menstrual blood loss. The total score is calculated by adding up the sum of all scores for the tampons or sanitary napkin used in the menstrual cycle. For tampons: 1 for lightly stained, 5 for moderately soiled and 10 for completely saturated tampons. For sanitary napkins: 1 for lightly stained, 5 for moderately soiled, and 20 for completely saturated pads. Clots were given a score of 1 for small and 5 for large clots. Abnormal PBLAC bleeding score greater than or equal to 100, which correlates with menorrhagia, defined as greater than 80 mL of menstrual blood loss. Normal bleeding is defined as a score of 75 or less. A score of 0 indicates amenorrhea, or absence of menstruation.
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
units on a scale | 15 [0 to 131] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Quality of Life Score Using the Short Form-12 (SF-12) Health Survey
Description: Quality of life (QoL) was measured by the SF-12 questionnaire. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. Physical and Mental Health Composite Scores are computed (combined, scored, and weighted) using the scores of the 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Improvement was defined as a change of ≥ 6 points.
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
units on a scale
  SF-12 Physical Scale | 54.2 (5.9) | 54.5 (4.2)
  SF-12 Mental Scale | 49.8 (10.0) | 53.8 (6.6)
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Comparison between the groups for the SF-12 Physical Scale; Test type: Superiority or Other; p = 0.82, t-test, 2 sided
Statistical Analysis 2: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Comparison between the groups for the SF-12 mental scale; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

3. Secondary Outcome: Quality of Life as Measured by the Menorrhagia Multi-Attribute Scale (MMAS )
Description: The MMAS questionnaire captures the subjective consequences of menorrhagia on six domains: practical difficulties; social life; psychological wellbeing; physical health; work routine; and family life. Each of the six domains has four statements that represent four levels of response. Respondents indicate the statement that best matches their feelings for each domain. The statement scores derive from a weighting of the domains and a weighting of the statements in level of severity by women in the original study. Scores range from 0 (worst possible state in all domains) to 100 (best possible state in all domains).
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
units on a scale | 100 [87.2 to 100.0] | 100 [100.0 to 100.0]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Hemoglobin at 12 Months
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
g/dL | 13.2 [12.5 to 13.8] | 13.4 [12.7 to 13.9]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Hemoglobin
Time Frame: baseline, 12 months
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
g/dL | 0.0 [-0.6 to 0.7] | 0.5 [0.0 to 2.2]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Ferritin at 12 Months
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
ug/L | 25.0 [17.0 to 33.0] | 26.5 [15.0 to 39.0]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Ferritin From Baseline
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
ug/L | 4.0 [-1.0 to 16.0] | 10.0 [4.0 to 22.0]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Direct Medical Costs
Description: Direct Medical Costs consisted of two categories: primarily hospital billed services, and primarily physician billed services. Primary hospital billed services were as defined by Medicare billing practice.
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
dollars
  Primarily hospital billed services | 1300 (1170) | 3494 (4006)
  Primarily physician billed services | 1601 (1576) | 1837 (1602)

9. Secondary Outcome: Indirect Medical Costs
Description: Indirect cost A refers to cost of sanitary products and lack of activity, indirect cost B refers to cost of sanitary products and reduced work days, and indirect cost C refers to cost of sanitary products, lack of activity, and reduced work days.
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
dollars
  Indirect costs A | 741 (1174) | 124 (403)
  Indirect costs B | 264 (467) | 27 (79)
  Indirect costs C | 968 (1534) | 138 (421)

10. Secondary Outcome: Bleeding Pattern at 12 Months
Description: The menstruation pattern of the subjects was evaluated. A bleeding episode was defined as any set of one or more bleeding days bounded at each end by two or more bleeding-free days. The bleeding pattern was analyzed using a 90 day reference period and divided into groups, (based on World Health Organization (WHO) classification of clinically important bleeding patterns). The groups are Amenorrhea (no bleeding during the reference period); Infrequent bleeding (fewer than 3 bleeding episodes); Irregular bleeding (between 3 and 5 episodes with less than 3 bleeding-free intervals of length 14 days or more); Prolonged bleeding (1 or more bleeding episodes lasting 14 days or more); Eumenorrhea "normal pattern" (none of the above patterns).
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
participants
  Amenorrhea | 5 | 16
  Irregular/Infrequent bleeding | 4 | 6
  Prolonged bleeding | 2 | 0
  Eumenorrhea | 8 | 9

11. Secondary Outcome: Pain at 12 Months as Measured by the Pain Visual Analog Scale (VAS)
Description: The pain VAS is a continuous scale comprised of a horizontal (HVAS) line, 100 mm in length. Possible scores range from 0 (no pain) to 100 (worst possible pain). The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
mm | 0.4 [0.0 to 3.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Medical Therapy vs Radiofrequency Endometrial Ablation; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Subject Satisfaction at 12 Months
Description: Subject satisfaction was ascertained by asking study participants to choose from one of four categories relating to their general satisfaction with treatment: totally satisfied, generally satisfied, acceptable improvement in symptoms, or unacceptable treatment.
Time Frame: Measured at 12 months following initial treatment
Population: Only subjects who completed the 12 month visit were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Number analyzed (Participants) | 19 | 31
participants
  Totally satisfied | 12 | 30
  Generally satisfied | 4 | 1
  Acceptable improvement | 2 | 0
  Unacceptable | 1 | 0

ADVERSE EVENTS:
Arm/Group | Medical Therapy | Radiofrequency Endometrial Ablation
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 12/33 | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Therapy (N=33) | Radiofrequency Endometrial Ablation (N=34)
Mild headache (General disorders) | 2 (2) | 0 (0)
Moderate headache (General disorders) | 4 (4) | 0 (0)
Gastrointestinal adverse events (Gastrointestinal disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Extremity edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0)
Increased blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes